CLINICAL TRIAL: NCT02899689
Title: Induction of Labor in Women With Unfavorable Cervix: Randomized Control Study Comparing Dilapan to Foley Bulb
Brief Title: Induction of Labor in Women With Unfavorable Cervix: Dilapan Versus Foley Bulb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Medicem International CR s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0272
Record Dates: First submitted 2016-08-31; First posted 2016-09-14 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2018-11

CONDITIONS: Pre-induction Dilation of Cervix
Keywords: Labor; Foley; Dilapan; Cervical Dilators; Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Foley Bulb Group (Active Comparator): Patients will have a Foley catheter inserted into the internal cervical os.
  Interventions: Device: Foley Catheter
- Dilapan Group (Experimental): Patients will have Dilapan sticks inserted into the internal cervical os.
  Interventions: Device: Dilapan

INTERVENTIONS:
Device: Dilapan — Using a sterile speculum, the cervix is visualized and cleaned with iodine. Under direct visualization, synthetic osmotic dilators (Dilapan-S) are inserted into the cervical canal with special attention to cross through the internal os.
  Other Names: Osmotic cervical dilator
  Arms: Dilapan Group
Device: Foley Catheter — Using a sterile speculum, the cervix is visualized and cleaned with iodine. Under direct visualization, a Foley catheter is inserted into the cervix and the balloon is filled with 60 ml of sterile 0.9% NaCl.
  Other Names: Foley Bulb
  Arms: Foley Bulb Group

SUMMARY:
Women undergoing mechanical cervical ripening for labor induction will be randomized to Dilapan-S® versus Foley bulb. The investigators hypothesized that osmotic cervical dilators (Dilapan-S®) are as effective as Foley bulb catheter in rates of vaginal delivery.

DETAILED DESCRIPTION:
Historically, mechanical methods were the first methods developed to ripen the cervix or to induce labor. Dilapan-S® a synthetic osmotic cervical dilator made of a patented hydrogel (AQUACRYL), works by stimulating the release of endogenous prostaglandins, which degrade collagen fibers and soften the cervix. Additionally, it dilates the cervix gradually and the effect is gentle as well as predictable. Recently, Dilapan-S® has been approved by the FDA as a mechanical dilator for cervical ripening. There are no data comparing this newly approved Dilapan-S® to the Foley catheter, the most commonly used mechanical dilator method. Therefore, The investigators propose a randomized controlled trial to determine the efficacy of Dilapan-S® compared with Foley catheter for cervical ripening before induction of labor in pregnant women greater than 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman scheduled for induction of labor.
* Age between 18 and 45 years.
* Understanding and capable to sign informed consent.
* Singleton pregnancy.
* Gestational age ≥ 37 0/7 weeks.
* Live fetus in cephalic presentation.
* Intact membranes.
* Pelvic exam (sterile vaginal exam) of less than or equal to 3cm and at most 60% effaced.

Exclusion Criteria:

* Iodine allergy.
* Active labor or oxytocin has been administered.
* Chorioamnionitis.
* Prior uterine or cervical surgery.
* Non reassuring fetal status requiring immediate delivery.
* Non-cephalic fetal presentation.
* Active vaginal bleeding from cervical os.
* Placenta previa.
* EFW > 5000 gm(non diabetic) or > 4500gm (diabetic).
* Other contraindication to vaginal delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 419 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - University of Texas, Galveston, Texas
  - UTMB Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2016 to February 2018 at UTMB Galveston
Period: Overall Study
Arm/Group | Foley Bulb Group | Dilapan Group
Started | 209 | 210
Completed | 209 | 208
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: These demographics includes all that were randomized. 2 participants withdrew consent in the dilapan group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Foley Bulb Group | Dilapan Group | Total
Number analyzed (Participants) | 209 | 210 | 419
Age, Continuous [Median (Full Range); unit: years] | 25 [18 to 44] | 25 [18 to 44] | 25 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 210 | 419
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 147 | 153 | 300
  Not Hispanic or Latino | 62 | 57 | 119
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 209 | 210 | 419
Gestational age [Median (Inter-Quartile Range); unit: weeks] | 39.0 [39 to 41] | 39 [37 to 41] | 39 [39 to 41]
Nulliparous [Count of Participants; unit: Participants] | 98 | 88 | 186
Bishop score at randomization [Median (Inter-Quartile Range); unit: scores on a scale] — The total score is calculated by assessing the following five components on manual vaginal examination by a trained professional: Cervical dilation in centimeters. Cervical effacement as a percentage. Cervical consistency by provider assessment/judgement.
  The highest possible score is 13 and the lowest possible score is 0. Bishop scores of less than 6 usually require that a cervical ripening method (pharmacologic or physical, such as a foley bulb) be used before other method
  scores on a scale | 3 [0 to 7] | 3 [0 to 8] | 3 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Vaginal Delivery
Description: Proportion of patients that delivered vaginal. (%)
Time Frame: Through study completion, an average of 1-2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
Participants | 169 | 159

2. Secondary Outcome: Time of Vaginal Delivery
Description: Delivery time frame in mins from cervical dilator insertion
Time Frame: 2-4 days
Measure: Median (Full Range); unit: minutes
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
minutes | 1291 [1203 to 1408] | 1441 [1343 to 1521]

3. Secondary Outcome: Time to Reach Active Stage of Labor as ≥ 6cm Cervical Dilation
Description: time from hospital admission to reach active stage of labor defined as ≥ 6 cm (mins)
Time Frame: 1-2 days
Measure: Median (Full Range); unit: minutes
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
minutes | 1011 [913 to 1074] | 1152 [1092 to 1205]

4. Secondary Outcome: Change in Bishop Scores
Description: Change in Bishop score from insertion to extraction of device. The total score is calculated by assessing the following five components on manual vaginal examination by a trained professional: Cervical dilation in centimeters. Cervical effacement as a percentage. Cervical consistency by provider assessment/judgement.
  The highest possible score is 13 and the lowest possible score is 0. Bishop scores of less than 6 usually require that a cervical ripening method (pharmacologic or physical, such as a foley bulb) be used before other method
Time Frame: 12-24 hrs
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
score on a scale | 3 [-3 to 9] | 2 [-2 to 11]

5. Secondary Outcome: Operative Deliveries
Description: Proportion of patients that delivered vaginal by forceps assistance or vacuum (%) assistance.
Time Frame: 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
Participants | 6 | 9

6. Secondary Outcome: Cesarean Deliveries
Description: Proportion of patients that delivered by cesarean (%).
Time Frame: 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
Participants | 50 | 39

7. Other Pre Specified Outcome: Analgesia Requirement
Description: Rate of women who require any analgesia used during insertion of the device
Time Frame: 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
Participants | 38 | 34

8. Other Pre Specified Outcome: Spontaneous Labor
Description: Rate of women underwent spontaneous labor (%)
Time Frame: 1-4 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pharmacological Agents for Labor Induction (Prostaglandins, Oxytocin)(%)
Description: Rate of women that required pharmacological cervical ripening agents (%) requirement (%)
Time Frame: 1-2 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Artificial Rupture of Membranes (AROM)
Description: Rate of women that had artificial rupture of membranes (AROM) (%)
Time Frame: 1-2 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Regional Anesthesia
Description: Rate of epidural/spinal analgesia (%)
Time Frame: 1-2 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Device Insertion Time
Description: Total duration of Dilapan-S® /Foley catheter insertion (mins)
Time Frame: 1-2 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
minutes | 666 (319) | 774.1 (295)

13. Other Pre Specified Outcome: Device Placement to Delivery Interval
Description: Interval from device placement to delivery (mins)
Time Frame: 1-4 days
Measure: Median (Full Range); unit: minutes
Arm/Group | Foley Bulb Group | Dilapan Group
Number analyzed (Participants) | 209 | 208
minutes | 1291 [1203 to 1408] | 1441 [1343 to 1521]

14. Other Pre Specified Outcome: Time After Mechanical Dilator
Description: Induction (Oxytocin/Prostaglandin initiation) to delivery interval (mins)
Time Frame: 1-2 days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Comparison of Labor Curves Between Both Interventions
Description: Labor curves using Kaplan Meier method comparing Dilapan-S to Foley balloon
Time Frame: 1-2 days
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Device Complications
Description: Rates of complications resulting from device insertion (%):
  Vaginal bleeding Vaso-vagal reaction from manipulation of the cervix Cervical laceration Retraction into the uterine cavity Rupture of membranes (Date/Time) Entrapment of the device Fragmentation of the device in the genital tract Rates of complications associated with cervical ripening(%) Uterine tachysystole/hypertonus Non reassuring fetal status Systemic adverse events (nausea, vomiting, diarrhea, fever, hypotension, tachycardia)
Time Frame: 1-2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of the trial: up to 2 weeks after discharge from hospital
Arm/Group | Foley Bulb Group | Dilapan Group
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/208
Serious Adverse Events (participants affected / at risk) | 2/209 | 0/208
Other Adverse Events (participants affected / at risk) | 0/209 | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foley Bulb Group (N=209) | Dilapan Group (N=208)
Serious Adverse event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin breakdown from mobility due to epidural. Unrelated to the study since device was already removed and epidural placed after the intervention (Foley balloon ) was removed. Occurred in the postpartum period
Motor vehicle collision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — 1 motor vehicle accident - occurred postpartum within 2 weeks of delivery. Resulted in prolonged hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02899689/Prot_SAP_000.pdf